CLINICAL TRIAL: NCT02647242
Title: Pilot Study on Feasibility and Safety of a Gait Auto-rehabilitation Program by Rhythmic Auditory Cueing Delivered by BeatHealth in Patients With Parkinson's Disease.
Brief Title: Proof of Concept BeatPark
Acronym: BEATPARK 2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion of the Last patient
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Université Montpellier (Other); University Ghent (Other); Tecnalia (Unknown); National University of Ireland, Maynooth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF 9193-4
Record Dates: First submitted 2016-01-05; First posted 2016-01-06 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with parkinson's disease (Experimental): Patients with parkinson's disease
  Interventions: Behavioral: Auto rehabilitation program of gait with Beat Health device.

INTERVENTIONS:
Behavioral: Auto rehabilitation program of gait with Beat Health device. — The auto-rehabilitation program will consist in an outside walk, during 5 sessions of 30 minutes per week during 4 weeks with the beatHealth device, delivering the optimal rythmic auditory cueing. The device will associate an Android smartphone, hold at the belt, connected by bluetooth to a headphone and to two sensors strapped to the ankles. The patient will transfer the data collected by BeatHealth to a secured website and will complete the agenda

SUMMARY:
Physical activity has demonstrated its beneficial effect on functional capabilities and quality of life in patients with PD. However, the daily physical activity remains limited in these patients. Rhythmic auditory cueing improves spatio-temporal gait parameters in patients with PD. The first results of BeatHealth studies have allowed us to identify the best musical stimulation to improve these parameters and the motivation of the patients.

The originality of this study is to propose a gait auto-rehabilitation program using BeatHealth device with optimal auditory cueing during four weeks in ecological conditions in PD.

Observance (utilization's time), safety (falls, pain, fatigability) and efficacy (gait parameters, balance, quality of life) will be evaluated.

DETAILED DESCRIPTION:
Objectives Main goal: To evaluate the observance of the use of BeatHealth device in gait auto-rehabilitation program in patients with PD.

Secondary objectives :

1. To evaluate safety by the number of falls
2. To evaluate tolerance by the evaluation of pain and fatigue
3. To evaluate the expected improvement on gate and quality of life essentialy
4. To identify predictive factors associated with a good response to the program
5. To evaluate the technical feasibility.

   Methods Design : prospective and descriptive study Population : 60 patients with PD Inclusion criteria : PD diagnosed according the international criteria form the United Kingdom Parkinson's Disease Society Brain Bank ; gait disorder identified by the neurologist or the rehabilitation doktor ; to be able to work 30 minutes consecutively and without technical support Non inclusion criteria : signs for atypical parkinsonism

   Main evaluation criteria:

   Percentage of time of use of the BeatHealth device compared to the prescribed schedule (30 minutes of walk, 5 times a week during four weeks : 10 hours for the complete study) .

   Secondary evaluation criteria :

   n°1 - Auto-evalation of the number of falls reported by the patient on a daily agenda before and during the rehabilitation program.

   n°2 - Auto-evalation of pain with a visual analogic scale on a daily agenda before and during the rehabilitation program.

   n°3 - (a) gait functional capabilities; (b) spatio-temporal parameters of gait; (c) motot severity of the disease(d) balance ; (e) quality of life ; (f) psychopathological evaluations (g) auditory-sensori-motor and timing capabilities (h) sleep.

   n°4 - Numbers of correct connections to the program, number of errors of manipulations, number of phone calls for help.

   Statistical analysis : In the randomized control study on 21 patients from Martin et al. (2015) evaluating a rehabilitation programm on rythmic auditory cueing by metronome in patients with PD wiht fall potential, program observance was 83% according to self evaluation by the patients. In our study , to estimate this percentage of about 80% with an accuracy of ± 10% (interval of 20%) with a confidance interval of 95, the number of subjects to include is 60.

   Main statistical analysis : in order to evaluate the observance of the BeatHealth device, the percentage of the time of use conpared to the prescribed time (10 hours in total)

   Program schedule :

   Number of visits : 3 Inclusion period : 7 months Follow-up : 2 weeks (from the inclusion to the beginning of the program) + 4 weeks (program) Calendar of the study : january 2016 - october 2016

   Content of the visites :

   V0=Inclusion / identification of the favorite musical genres of the patient / Explanation and delivery of the agenda.

   V1=
   * Evalutation criteria
   * Information and training to the BeatHealth device use (sensors, smartphone use, connexion to the cloud for the transfer of the results)
   * Operating instructions delivery
   * Explanation of the rehabilitation program (number of sessions, duration, place…)
   * Communication of the contact details of the maintenance operator V2= identical to V1 (except for predictive factors).

   Description of the intervention The auto-rehabilitation program will consist in an outside walk, during 5 sessions of 30 minutes per week during 4 weeks with the beatHealth device, delivering the optimal rythmic auditory cueing. The device will associate an Android smartphone, hold at the belt, connected by bluetooth to a headphone and to two sensors strapped to the ankles. The patient will transfer the data collected by BeatHealth to a secured website and will complete the agenda

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease confirmed by the United Kingdom Parkinson's Disease Society Brain Bank's criteria (Gibb and Lees, 1988; Hughes et al., 1992)
* Gait disorder confirmed by a neurologist
* Ability to walk more than 30 minutes without any device as a stick or a walker
* Stability of the dopaminergic treatment

Exclusion Criteria:

* Pregnancy
* Hearing problems
* Other neurological disease affecting gait other than PD
* Other gait disorder whetever the etiology (orthopedic, rheumatologic….)
* Uncompensated heart or respiratory failure excluding possibility of intensiv rehabilitation.
* Arguments for atypical parkinsonism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
Percentage of time of use of the BeatHealth device compared to the prescribed schedule | 4 weeks
  measured automatically by Beathealth device

SECONDARY OUTCOMES:
Auto-evalation of the number of falls reported by the patient on a daily agenda | 4 weeks
  self reported in a diary

REFERENCES:
- [Derived] Cochen De Cock V, Dotov D, Damm L, Lacombe S, Ihalainen P, Picot MC, Galtier F, Lebrun C, Giordano A, Driss V, Geny C, Garzo A, Hernandez E, Van Dyck E, Leman M, Villing R, Bardy BG, Dalla Bella S. BeatWalk: Personalized Music-Based Gait Rehabilitation in Parkinson's Disease. Front Psychol. 2021 Apr 26;12:655121. doi: 10.3389/fpsyg.2021.655121. eCollection 2021. PMID 33981279